CLINICAL TRIAL: NCT03972228
Title: Pilot Study of Microdevice for Evaluating Drug Response in Site in Lung Lesions
Brief Title: Microdevice for Evaluating Drug Response in Site in Lung Lesions
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oliver Jonas (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Oliver Jonas, Co-Investigator, Division of Radiology, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017P002401
Record Dates: First submitted 2019-03-25; First posted 2019-06-03 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Lung Tumor; Lung Cancer
Keywords: microdevice; chemotherapy; lung lesions
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Microdevice Intervention (Experimental): The intervention to be administered is the placement of the microdevice containing 19 FDA-approved drugs into the lung lesion and the device's subsequent surgical resection. All study subjects will receive this same intervention; there is only one arm.
  Interventions: Combination Product: Microdevice loaded with 19 chemotherapeutic agents

INTERVENTIONS:
Combination Product: Microdevice loaded with 19 chemotherapeutic agents — The microdevice containing 19 FDA-approved chemotherapeutic agents will be placed in the suspected tumor tissue at the time of surgical resection. Multiple chemotherapeutic agents will passively diffuse into local, confined regions (several microns) of the surrounding microenvironment. The agents are released at approximately one millionth of a systemic dose. The device(s) will be removed for analysis at the time of resection, which will be performed for clinical indications independent of enrollment in this study.

SUMMARY:
This is a pilot study for placement of a tiny microdevice into lung tumors to more precisely predict tumor-specific drug sensitivity, and to help inform systemic therapeutic decisions. The microdevice will provide a novel technique for interrogating human lung tumor tissue in situ, and will uniquely facilitate assessment of response to multiple drugs simultaneously. This will not only increase the specificity of a particular participant's chosen systemic therapy, it will also augment the speed and efficiency with which investigators are able to make clinical decisions regarding choice of therapy.

DETAILED DESCRIPTION:
The initial aims in this pilot study will focus on the safety and feasibility of microdevice placement and retrieval in participants with suspicious lung lesions. The microdevice, which is 5.5 mm in length and approximately 750 µm in diameter (i.e., comparable in size and shape to commonly used fiducial markers), will be placed in the suspected tumor tissue at the time of surgical resection. Multiple agents will passively diffuse into local, confined regions (several microns) of the surrounding microenvironment. The agents are released at approximately one millionth of a systemic dose. The device(s) will be removed for analysis at the time of resection, which will be performed for clinical indications independent of enrollment in this study. The investigators will collect data regarding the safety and feasibility of the placement and retrieval of the microdevices, and perform detailed tissue analysis of drug response. Investigators hope to compile preliminary data regarding correlations between in situ drug response and the genetic and histopathologic features of tumors, systemic treatment response, and ultimately, clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a suspicious lung lesion for which surgery is indicated for either diagnostic or therapeutic purposes, as determined by the treating thoracic surgeon
* Masses with a minimum longest dimension of 1 cm
* 18 years of age or older
* Documented, signed, dated informed consent for both the surgical resection as well as the proposed research study obtained prior to any procedures

Exclusion Criteria:

* Subjects who do not wish to undergo surgical resection, or those who are high-risk or not candidates for surgical resection in the opinion of the treating surgeon
* Women of childbearing potential without a negative pregnancy test; or women who are lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and feasibility) related to the placement and removal of the microdevice. | 5 years
  Safety will be measured quantitatively by the number of participants with treatment-related adverse events.
Number of histopathology analyses and interpretations for drugs eluted from microdevice reservoirs into resected lung lesion tissue. | 5 years
  Feasibility will be based on the ability to retrieve the device with sufficient tissue, of sufficient quality, for downstream histopathology analysis and interpretation of the device reservoirs.

SECONDARY OUTCOMES:
Stratification of local tumoral cellular responses to various agents and combinations of agents released from the microdevice reservoirs. | 5 years
  This initial proof-of-concept pilot study will gauge the ability of using the microdevice to predict tumor drug response, allowing a stratified systemic treatment to prioritize those agents inducing the greatest anti-tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: Yolonda L Colson, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Tsai LL, Phillips WW, Hung YP, Dominas C, Deans K, Ahn S, Ferland B, Weiss K, Lanuti M, Auchincloss H, Schumacher L, Jonas O, Colson YL. First-in-Human Intrathoracic Implantation of Multidrug-Eluting Microdevices for In Situ Chemotherapeutic Sensitivity Testing as Proof of Concept in Nonsmall Cell Lung Cancer. Ann Surg. 2023 May 1;277(5):e1143-e1149. doi: 10.1097/SLA.0000000000005385. Epub 2023 Apr 6. PMID 35129472